CLINICAL TRIAL: NCT00801359
Title: Comparison of Corneal Changes After Phacoemulsification Using BSSPlus Versus Lactated Ringer's Irrigating Solution
Brief Title: BSSPlus Versus Lactated Ringer's for Phacoemulsification
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Rodrigo Jorge, University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 8657/2007
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-12

CONDITIONS: Cataract
Keywords: cataract; phacoemulsification; irrigation solution; endothelial cell density; corneal thickness
MeSH Terms: conditions — Cataract | interventions — Phacoemulsification; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BSSplus (Active Comparator)
  Interventions: Procedure: Phacoemulsification; Drug: BSSPlus solution
- Ringer (Experimental)
  Interventions: Procedure: Phacoemulsification; Drug: Lactated Ringer's solution

INTERVENTIONS:
Procedure: Phacoemulsification
Drug: BSSPlus solution
  Arms: BSSplus
Drug: Lactated Ringer's solution
  Arms: Ringer

SUMMARY:
Two intraocular irrigating solutions (BSSPlus versus Lactated Ringer's) are compared in this prospective, randomized, masked trial to investigate for differences in preservation of corneal integrity after phacoemulsification cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with senile cataract
* Visual acuity between 20/400 and 20/40

Exclusion Criteria:

* Presence of corneal opacity
* Presence of corneal disease
* Traumatic, toxic, hereditary (congenital)and complicated cataracts(uveitis)
* Anterior chamber cells or flare detected before surgery
* Previous ocular surgery
* Any condition which may affect documentation or follow-up

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2008-01; Primary Completion 2008-08 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
endothelial cell density | baseline and at 1, 8, 15, 30 and 60 days postoperatively
central corneal thickness | baseline and at 1, 8, 15, 30 and 60 days postoperatively

SECONDARY OUTCOMES:
number of anterior chamber cells and flare grade | baseline and at 1, 8, 15, 30 and 60 days postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto; Centro Avançado de Retina e Catarata, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Background] Puckett TR, Peele KA, Howard RS, Kramer KK. Intraocular irrigating solutions. A randomized clinical trial of balanced salt solution plus and dextrose bicarbonate lactated Ringer's solution. Ophthalmology. 1995 Feb;102(2):291-6. doi: 10.1016/s0161-6420(95)31026-3. PMID 7862416
- [Background] McCarey BE, Polack FM, Marshall W. The phacoemulsification procedure. I. The effect of intraocular irrigating solutions on the corneal endothelium. Invest Ophthalmol. 1976 Jun;15(6):449-57. PMID 931689
- [Background] Joussen AM, Barth U, Cubuk H, Koch H. Effect of irrigating solution and irrigation temperature on the cornea and pupil during phacoemulsification. J Cataract Refract Surg. 2000 Mar;26(3):392-7. doi: 10.1016/s0886-3350(99)00470-8. PMID 10713235
- [Background] Kaye GI, Mishima S, Cole JD, Kaye NW. Studies on the cornea. VII. Effects of perfusion with a Ca++-free medium on the corneal endothelium. Invest Ophthalmol. 1968 Feb;7(1):53-66. No abstract available. PMID 5636786
- [Background] Rosenfeld SI, Waltman SR, Olk RJ, Gordon M. Comparison of intraocular irrigating solutions in pars plana vitrectomy. Ophthalmology. 1986 Jan;93(1):109-15. doi: 10.1016/s0161-6420(86)33790-4. PMID 3513079